CLINICAL TRIAL: NCT04035759
Title: Positive Affect Promotion to Empower Optimal Adherence to HIV Therapy (Project APPEAL)
Brief Title: Positive Affect Promotion to Empower Optimal Adherence to HIV Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: State University of New York - Downstate Medical Center (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Tracey Wilson, Professor, Community Health Sciences, State University of New York - Downstate Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1259781; R21NR018348 (NIH)
Record Dates: First submitted 2019-07-23; First posted 2019-07-29 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APPEAL Program (Experimental): Participants receive the APPEAL program, consisting of three one-on-one sessions, each lasting approximately one hour, and spaced one month apart. Sessions are designed to promote positive affect. Participants receive optional weekly check-ins to support behavior change efforts. All participants continue to receive standard of care.
  Interventions: Behavioral: APPEAL
- Standard of care (No Intervention): Participants receive standard of care.

INTERVENTIONS:
Behavioral: APPEAL — Three-session, individually administered program, with sessions spaced monthly. Optional weekly contacts with participants to support engagement in program exercises/activities.
  Arms: APPEAL Program

SUMMARY:
This study assesses the feasibility and acceptability of the APPEAL program, a 3-session intervention designed to promote positive affect among men and women living with HIV infection. Forty participants will be randomly assigned to receive the APPEAL program, and another 40 will receive standard of care. All participants will complete self-reported assessments at baseline and at 3 and 6 months, and will have their HIV antiretroviral medication adherence monitored as part of study participation.

DETAILED DESCRIPTION:
There is strong reason to expand the scope of current adherence programs to include consideration of a group of health protective variables known as 'psychosocial assets'. These assets include cognitive factors, such as optimism, emotional factors, such as positive affect, and positive social relationships. Increased psychosocial assets such as positive affect are associated with reduced morbidity and mortality, slower slower HIV progression, and reduced burden of depression symptoms. However, there has been limited translation of positive affect interventions to support patient self-management. In this study, we extend previous research on positive affect and adherence through the APPEAL program. The Affect, Promoting Positive Engagement, and Adherence for Life (APPEAL) program is an intervention that combines positive affect approaches to promote adherence in patients who have suboptimal adherence. We seek to implement the program, assess its feasibility, and describe associations with theoretically derived mechanisms of change, including positive affect.

ELIGIBILITY:
Inclusion Criteria:

* Receiving HIV care at site of recruitment
* Prescribed an HIV antiretroviral regimen
* HIV RNA viral load less than 200 copies/mL in last six months

Exclusion Criteria:

* Unable to communicate in English
* Prior participation in formative components of the study
* Plans to move outside of New York City in next six months
* Has cognitive impairment that would limit ability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment approaches | Baseline to 6 months
  The percentage of eligible individuals consented and randomized
Feasibility of retention methods | Baseline to 3 months
  The percentage of enrolled individuals who complete baseline, three-month, and six-month self-report evaluation measures
Acceptability of intervention | Baseline to 6 months
  The percentage of individuals in the intervention condition who complete all three sessions
Changes in the proposed mechanistic target of positive and negative emotions, assessed using the Positive and Negative Affect Scale (PANAS) | Baseline, 3 months, 6 months
  The PANAS is a 20 item measure which assesses emotions utilizing 5 response options for each question, ranging in value from 1 to 5. PANAS includes two 10-item subscales: positive affect and negative affect. Positive affect and negative affect items are summed separately, with each subscale ranging from 10 to 50. Higher scores for positive affect subscale indicate higher levels of positive affect and lower scores for negative affect items indicate lower levels of negative affect

SECONDARY OUTCOMES:
Measurement properties (range, missingness, reliability) and mean scores with standard deviations for the Modified Differential Emotions Scale (MDES). | Baseline, 3 months, 6 months
  The MDES is a 20 item measure which assesses emotions utilizing 5 response options for each question, ranging in value from 0 to 4. MDES includes two 10-item subscales: positive affect and negative affect. Positive affect and negative affect items are summed separately, and each is divided by 10, with each subscale ranging from 0 to 4. Higher score for each subscale indicate greater frequency of experiencing positive or negative emotions.
Measurement properties (range, missingness, reliability) and mean scores with standard deviations for the Drug Abuse Screening Test (DAST 10) | Baseline, 3 months, 6 months
  The DAST 10 is a 10 item screen for drug abuse. It includes 10 items, each response with a 0 or 1. Items are summed, with a range of responses from 0 to 10. Higher scores indicate greater negative consequences of drug abuse.
Measurement properties (range, missingness, reliability) and mean scores with standard deviations for the Perceived Stress Scale (PSS4) | Baseline, 3 months, 6 months
  The PSS4 measures perceived stress. Each of the 4 items has five possible response options, ranging from 0 to 4. The resulting summed scale can range from 0 to 16, with higher scores indicating greater stress.
Measurement properties (range, missingness, reliability) and mean scores with standard deviations for the Coping Strategies Inventory, Short Form (CSISF) | Baseline, 3 months, 6 months
  The CSISF is a 16 item scale assessing approaches to coping with stressors. Each of the items has 5 potential response options, ranging from 1 to 5, and items are grouped into four 4-item subscales. Items within each subscale are summed, resulting in a subscale range from 4 to 20. Higher scores on each of the subscales, focused on 1) Problem-Focused Engagement, (2) Problem-Focused Disengagement, (3) Emotion-Focused Engagement, and (4) Emotion-Focused Disengagement, indicates greater frequency of use of that particular coping strategy.
Measurement properties (range, missingness, reliability) and mean scores with standard deviations for the Revised Life Orientation Test (LOT-R) | Baseline, 3 months, 6 months
  The LOT-R is a 6-item measure of generalized optimism versus pessimism. For each of the items there are 5 response options ranging from 0 to 4. Items are summed with a scale range of 0 to 24, and with higher scores indicating greater optimism.
Measurement properties (range, missingness, reliability) and mean scores with standard deviations for the Patient Health Questionnaire-8 item (PHQ8) | Baseline, 3 months, 6 months
  The PHQ8 is an 8-item measure assessing burden of depression symptoms. Each item has 4 response options ranging from 0 to 3; items are summed with a resulting scale range of 0 to 24. Higher scores suggest greater risk for depression.
Measurement properties (range, missingness, reliability) and mean scores with standard deviations for the Alcohol Use Disorders Identification Test - Concise (AUDIT-C) | Baseline, 3 months, 6 months
  The AUDIT-C is a 3-item measure assessing risk for alcohol use disorder. Each item has 4 response options ranging from 0 to 4, and items are summed with a resulting range from 0 to 12. In men, a score of 4 or more is considered positive for an alcohol use disorder; in women, a score of 3 or more is considered positive.
Frequency of endorsement of stressful life events utilizing a modification of the Crisis in Family Systems (CRYSIS) | Baseline, 3 months, 6 months
  An adapted version of the CRISYS checklist is being utilized, based on formative feedback on the scale. The adapted measure lists thirty-four events, with a 0 indicating no experience and a 1 indicating an experience. The checklist can range from 0 to 34 possible events.
Self-reported values of percent adherence | Baseline, 3 months, 6 months
  Single item asking over past 30 days how often medication was taken as prescribed. Four response options available: 100%, 95-99% 75-94%, less than 75%
Self-reported adherence with medication taking instructions | Baseline, 3 months, 6 months
  Single item asking over past 30 days how good of a job did participant do at take medication in the way that they are supposed to. Six response options available: Very poor, poor, fair, good, very good, excellent
Self-reported adherence missed doses of medication | Baseline, 3 months, 6 months
  Single item asking number of days in the past 30 days that participant missed at least one dose of medication
Feasibility of electronic medication adherence | Baseline through 6 months
  Proportion of participants who utilize Wisepill throughout study participation
HIV RNA viral load | Baseline through 6 months
  Chart review will be conducted to assess HIV RNA viral load
Retention in care | Baseline through six months
  Chart review will be conducted to assess kept and missed study visits

CONTACTS AND LOCATIONS:
Overall Officials: Tracey Wilson, PhD, Principal Investigator — SUNY Downstate Health Sciences University
Locations (1):
- SUNY Downstate Health Sciences University, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Raw, de-identified data and codebook related to primary outcomes will be made available on Open Science Framework.
  Wilson, T. (2019, July 21). Positive Affect Promotion to Empower Optimal Adherence to HIV Therapy. Retrieved from osf.io/s7ve9
Time Frame: Data will become available upon completion of publication of outcomes paper associated with the study. Data will be made available for three years following publication.
Access Criteria: Principal Investigator wil grant permission upon request
URL: http://osf.io/s7ve9

REFERENCES:
- [Derived] Wilson TE, Massiah C, Radigan R, DeHovitz J, Govindarajulu US, Holman S, Melendez M, Yusuff J, Taylor T. The positive affect, promoting Positive Engagement, and Adherence for Life (APPEAL) feasibility trial: Design and rationale. Health Psychol. 2020 Sep;39(9):767-775. doi: 10.1037/hea0000880. PMID 32833478